CLINICAL TRIAL: NCT00327041
Title: Pilot Study Investigating the Use of a Variety of Assays to Detect Individual Response to Antiplatelet Therapy
Brief Title: Monitoring Response to Antiplatelet Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Other Study IDs: rgoodtrial001
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-05-17 (Estimated); Status verified 2006-05

CONDITIONS: Coronary Stenosis; Coronary Thrombosis; Angioplasty, Balloon
Keywords: Aspirin; Clopidogrel; Balloon Angioplasty; Coronary Thrombosis
MeSH Terms: conditions — Coronary Stenosis; Coronary Thrombosis

SUMMARY:
Antiplatelet therapy plays a key role in the prevention of complications related to coronary angioplasty and stenting (PCI) including procedure related myocardial damage. Aspirin and clopidogrel are now universally prescribed in patients undergoing these procedures. However, loading and maintenance doses have not been established and variation in individual response is emerging. New tests to assess the effects of these drugs are being developed but have yet to be incorporated into routine clinical practice. We will assess the effects of aspirin and clopidogrel in a consecutive series of patients undergoing angioplasty using new assays which can be carried out at the bedside. We will compare the results with alternative laboratory based tests and look for an association between the results, peri-procedural myocardial necrosis and subsequent cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-80 undergoing intended PCI for conventional indications. Informed written consent.

Exclusion Criteria:

Administration of GPIIbIIIa therapy prior to PCI, Oral anticoagulation, ticlopidine, dipyridamole, NSAID therapy, Pregnancy, Troponin I >0.2mcg/l on day of procedure, Chest pain in the 24 hrs prior to PCI. Anaemia (Hb<10g/dl). Platelet Count <150 or >450 x10^9/l, Personal or family history of bleeding disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Oldroyd, MBChB, MD, FRCP, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Western Infirmary, Glasgow, Scotland, United Kingdom